CLINICAL TRIAL: NCT07302113
Title: Promoting Health-Related Quality of Life in Pediatric Lupus Patients: Development and Implementation of a Tailored Brain Health Intervention
Brief Title: Complete Cognitive Intervention for cSLE
Acronym: CCIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Knight (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor-Investigator, Andrea Knight, Clinical Investigator, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3413
Record Dates: First submitted 2025-11-18; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lupus
Keywords: lupus; psychological intervention; adolescent; cognitive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOPS (Experimental)
  Interventions: Behavioral: Lupus Teen Online Problem Solving program

INTERVENTIONS:
Behavioral: Lupus Teen Online Problem Solving program — The Lupus Teen Online Problem Solving program is a brain health intervention developed to meet the needs of youth with childhood-onset lupus. The original Teen Online Problem Solving Program (TOPS) was developed for use with families impacted by traumatic brain injury. The Lupus Teen Online Problem Solving program is based on TOPS, with modifications to maximize relevance and accessibility. The intervention is a 10 session, evidence-based telehealth program providing training in problem-solving, emotion regulation, and communication skills in a one-to-one therapist-mediated design.

SUMMARY:
This project will work closely with patients to design and test a new program that supports brain health in children and youth with childhood-onset lupus (cSLE). The investigators will see how practical and helpful the program is for patients.

DETAILED DESCRIPTION:
The proposed project will use a patient-informed participatory action approach to develop and assess preliminary feasibility and acceptability of an intervention tailored to address the specific brain health needs of cSLE patients.

ELIGIBILITY:
Inclusion Criteria:

* Receive subject-informed consent;
* Have a current diagnosis of cSLE that meets the 1997 American College of Rheumatology (ACR) or System Lupus International Collaborating Clinics (SLICC) classification criteria
* Aged 13-18 years old

Exclusion Criteria:

* Conditions that significantly affect cognition (e.g., intellectual disability diagnosis, active psychosis), hearing loss or vision problems precluding participation in group
* Non-English speaking
* Lack of access to technology that would allow them to participate in the virtual intervention (e.g., phone, tablet, computer, etc.)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited | 1 year
  Feasibility will be assessed by rates of participant recruitment.
Number of intervention sessions attended | through study completion, an average of 1 year
  Feasibility will be assessed by rates of participant session attendance.
Number of participants completing the intervention | through study completion, an average of 1 year
  Feasibility will be assessed by rates of participant intervention completion.
Acceptability ratings | 0-2 weeks post-intervention
  Participant acceptability will be determined ratings of their satisfaction with aspects of the program on a brief survey using 5-point Likert scales (ranging from "dissatisfied" to "extremely satisfied").
Qualitative feedback on feasibility and acceptability of the intervention | 0-2 weeks post-intervention
  Semi- structured interviews administered to participants post-intervention will also assess intervention feasibility and acceptability.

SECONDARY OUTCOMES:
Depressive symptoms | Baseline and 10 weeks
  The 21-item Beck Depression Inventory-II will be used to assess depressive symptoms. Minimum possible total score of 0 and a maximum possible total score of 63. Higher scores means worse.
Anxiety symptoms | Baseline and 10 weeks
  The 41-item Screen for Child Anxiety Related Disorders self-report form will be used to assess anxiety symptoms. Minimum total score 0 and the maximum total score 82. Higher means worse.
Executive function | Baseline and 10 weeks
  The self-report Behavior Rating Inventory of Executive Function, Second Edition will be used to assess executive functioning skills, defined as a set of higher-level cognitive skills that enable problem-solving and goal-directed behaviour.
Self-efficacy | Baseline and 10 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions scale will be used to measure self-efficacy, defined as an individual's belief in their capacity to act in the ways necessary to reach specific goals. Scores range 4-20 with higher scores meaning better efiicacy.
Social engagement | Baseline and 10 weeks
  The PROMIS Social Role Participation will be used to assess participants' social engagement. Scale is 20-80. Higher score is better.
Medication adherence | Baseline and 10 weeks
  The Medication Adherence Self-Report Inventory will be used to measure adherence to medication. 0-100% scale with higher meaning better medication adherence.
Health-related quality of life | Baseline and 10 weeks
  The Pediatric Quality of Life Inventory (PedsQL) will be used to assess participants' health-related quality of life, including aspects of physical functioning, emotional functioning, social functioning, and school functioning. 0-100 range with higher being better.

CONTACTS AND LOCATIONS:
Overall Officials: Busi Zapparoli, PhD, Principal Investigator — The Hospital for Sick Children; Andrea Knight, MD, MSCE, Principal Investigator — The Hospital for Sick Children

IPD SHARING:
Plan to Share IPD: Yes
Data will shared upon request and approval of the study plan by the PI, and when the appropriate data use agreement and ethical protocols are in place.